CLINICAL TRIAL: NCT06365242
Title: Direct Oral Anticoagulants and Management of Blleding Following Dental Extractions. A Prospective Cohort Study.
Acronym: DOACS_1
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonio Barone, Full Professor of Oral Surgery and Implantology, Principal Investigator, University of Pisa
Other Study IDs: DOACS1_2024
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Hemorrhage
Keywords: Direct Oral Anticoagulants; oral Surgical Procedure; Post-operative complications
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DOACs treated patients: Patients treated with DOACs undergoing oral extractions

SUMMARY:
Evaluation of DOACs treatment on post-extraction bleeding

DETAILED DESCRIPTION:
Consecutive patients requiring at least one dental extraction were enrolled. DOACs regimen was either maintained or suspended. Patients were classified in subgroups depending on the number of teeth extracted per procedure (≤ 3 or > 3), the need for flap raising and the performance of osteotomy. Bleeding was recorded intraoperatively, perioperatively at 20, 40, 60 and 80 minutes after the procedure, and in the first seven days post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* patients under pharmacological treatment with DOACs
* patients requiring at least one dental extraction
* patients willing to take part in the study and to sign informed consent

Exclusion Criteria:

* patients below 18 years of age
* patients treated with antiplatelet therapy or vitamin K antagonists
* patients presenting with an International Normalized Ratio (INR) >3.0
* patients suffering from congenital or acquired coagulopathies (e.g. haemophilia, coagulation factors deficiency, von Willebrand disease, thrombocytopenia, cirrhosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to the Unit of Dentistry and Oral Surgery for dental extraction between 2021 and 2023 were enrolled in this study. All the study participants signed an informed consent form to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Peri-operative hemorrhage | 20 minutes to 80 minutes
  Evaluation of early post-operative hemorrhage classified as absent, mild, oozing, moderate, and severe.
Post-operative bleeding | day 1 to 7 post-operatively
  Evaluation of post-operative bleeding classified as absent, mild, oozing, moderate, and severe.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Barone, Principal Investigator — University of Pisa
Locations (1):
- U.O. Odontostomatologia e Chirurgia del Cavo Orale, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available as aggregate and anonymous data for sceintific publication purposes.

REFERENCES:
- [Result] Lee JY, Park SH, Kim DM, Ko KA, Park JY, Lee JS, Jung UW, Cha JK. Risk of post-operative bleeding after dentoalveolar surgery in patients taking anticoagulants: a cohort study using the common data model. Sci Rep. 2024 Apr 2;14(1):7787. doi: 10.1038/s41598-024-57881-7. PMID 38565933
- [Result] Darwish G. The Effect of Direct Oral Anticoagulant Therapy (DOACs) on oral surgical procedures: a systematic review. BMC Oral Health. 2023 Oct 11;23(1):743. doi: 10.1186/s12903-023-03427-8. PMID 37821865
- [Result] Lababidi E, Breik O, Savage J, Engelbrecht H, Kumar R, Crossley CW. Assessing an oral surgery specific protocol for patients on direct oral anticoagulants: a retrospective controlled cohort study. Int J Oral Maxillofac Surg. 2018 Jul;47(7):940-946. doi: 10.1016/j.ijom.2018.03.009. Epub 2018 Apr 10. PMID 29653869
- [Result] Cocero N, Basso M, Grosso S, Carossa S. Direct Oral Anticoagulants and Medical Comorbidities in Patients Needing Dental Extractions: Management of the Risk of Bleeding. J Oral Maxillofac Surg. 2019 Mar;77(3):463-470. doi: 10.1016/j.joms.2018.09.024. Epub 2018 Sep 26. PMID 30347201
- [Result] Hiroshi I, Natsuko SY, Yutaka I, Masayori S, Hiroyuki N, Hirohisa I. Frequency of hemorrhage after tooth extraction in patients treated with a direct oral anticoagulant: A multicenter cross-sectional study. PLoS One. 2022 Apr 7;17(4):e0266011. doi: 10.1371/journal.pone.0266011. eCollection 2022. PMID 35390010
- [Result] Patel JP, Woolcombe SA, Patel RK, Obisesan O, Roberts LN, Bryant C, Arya R. Managing direct oral anticoagulants in patients undergoing dentoalveolar surgery. Br Dent J. 2017 Feb 24;222(4):245-249. doi: 10.1038/sj.bdj.2017.165. PMID 28232717
- [Result] Cabbar F, Cabbar AT, Cosansu K, Cekirdekci EI. Effects of Direct Oral Anticoagulants on Quality of Life During Periprocedural Management for Dental Extractions. J Oral Maxillofac Surg. 2019 May;77(5):904-911. doi: 10.1016/j.joms.2018.11.032. Epub 2018 Dec 12. PMID 30611688
- [Result] Johnston S. An evidence summary of the management of patients taking direct oral anticoagulants (DOACs) undergoing dental surgery. Int J Oral Maxillofac Surg. 2016 May;45(5):618-30. doi: 10.1016/j.ijom.2015.12.010. Epub 2016 Jan 7. PMID 26774397
- [Result] Mauprivez C, Khonsari RH, Razouk O, Goudot P, Lesclous P, Descroix V. Management of dental extraction in patients undergoing anticoagulant oral direct treatment: a pilot study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2016 Nov;122(5):e146-e155. doi: 10.1016/j.oooo.2016.06.003. Epub 2016 Jun 22. PMID 27554378